CLINICAL TRIAL: NCT01630161
Title: Smoking Relapse-Prevention Intervention for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCC-16458; 5R01CA154596-02 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
Keywords: relapse; prevention; smoking; habit; Forever Free
MeSH Terms: conditions — Smoking Cessation; Recurrence; Smoking; Habits

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to the Usual Care condition will receive standard care following recruitment.
  Interventions: Behavioral: Usual Care
- Relapse-Prevention Intervention (Active Comparator): Participants randomized to the Smoking Relapse Prevention for Cancer Patients (SRP-CaP) intervention will receive standard care plus our self-help smoking-relapse prevention materials.
  Interventions: Behavioral: Smoking Relapse Prevention for Cancer Patients (SRP-CaP)

INTERVENTIONS:
Behavioral: Usual Care — Standard care includes routine assessment of smoking behavior and brief clinical intervention. Smoking counseling for all participants in the current study will be completed by a Certified Tobacco Treatment Specialist consisting consists of brief counseling (<15 minutes) based on the 5 A's Clinical Practice Guidelines; Ask about tobacco use, Advise to quit, Assess willingness to make a quit attempt, Assist in quit attempt, Arrange for follow-up (Fiore et al., 2008). Patients receive information for local and state smoking resources (e.g., Quitline), pharmacotherapy options, and if interested, assistance with obtaining a prescription for pharmacotherapy. Follow-up with patients occurs at 2-weeks, only among those who are prescribed smoking medications (i.e., Varenicline, Bupropion).
  Arms: Usual Care
Behavioral: Smoking Relapse Prevention for Cancer Patients (SRP-CaP) — The proposed multimodal intervention consists of a series of easy-to-read relapse prevention booklets (Forever Free) that have shown to be efficacious with a general smoking population (Brandon et al., 2000; 2004), and digital video disk (DVD) customized to the needs of cancer patients (to be developed in Year One).
  Arms: Relapse-Prevention Intervention

SUMMARY:
The purpose of this study is to test different ways to help cancer patients maintain their smoking abstinence. Participants may receive educational materials as part of the study.

DETAILED DESCRIPTION:
This study involves participation at four distinct time points over a one-year period.

* Baseline assessment
* 2-month follow-up telephone call
* 6-month follow-up telephone call
* 12-month follow-up telephone call

ELIGIBILITY:
Inclusion Criteria:

* Have smoked at least 10 cigarettes per day for at least one year prior to cancer diagnosis
* Able to read and write English
* Able to give informed consent
* Have quit smoking after receiving their cancer diagnosis
* Have not quit greater than 3 months prior

Exclusion Criteria:

* Individuals who have been abstinent for greater than 3 months are not included because they are less likely to relapse. A quit will be defined as self-reported no smoking for 24 hours. Individuals with metastatic disease will be excluded because participation in the study might be burdensome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Relapse at 6 Months | 6 Months
  Number of participants with smoking relapse at 6 months follow-up for each treatment arm.
Number of Participants with Relapse at 12 Months | 12 Months
  Number of participants with smoking relapse at 12 months for each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Vani Simmons, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States